CLINICAL TRIAL: NCT03225963
Title: Application of Proteome Profiler Antibody Arrays to Find Angiogenetic Predictors in Glioma Paitents.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE15180B
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Glioblastoma Multiforme; Angiogenesis
Keywords: Glioblastoma; Bevacizumab
MeSH Terms: conditions — Glioblastoma | interventions — Chemoradiotherapy; Temozolomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA of peripheral mononulcear cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Chemoradiation with temozolomide

SUMMARY:
Bevacizumab has become the standard of care of recurrent glioblastoma based on promising clinical trial results with with response rates up to 50% and progression-free survival up to 9 months. In our study, we set to find the serum angiogenesis biomarkers of bevacizumab response.

DETAILED DESCRIPTION:
Pre-chemoradiation and post-chemoradiation peripheral blood will be obtained to see if there are some angiogenesis biomarker available for prediction of bevacizumab response later.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 20 year old.
* Glioblastoma patients who will receive chemoradiation treatment.

Exclusion Criteria:

* None

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obtain peripheral blood pre-chemotherapy, mid-chemoradition and post-chemoraidtion
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Response of bevacizumab therapy. | 3 months after bevacizumab therapy
  Base on the image after bevacizumab therapy (after recurrence)

CONTACTS AND LOCATIONS:
Overall Officials: Weir Chiang You, M.D. Ph.D., Study Chair — The Institutional Review Board of Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Lamszus K, Ulbricht U, Matschke J, Brockmann MA, Fillbrandt R, Westphal M. Levels of soluble vascular endothelial growth factor (VEGF) receptor 1 in astrocytic tumors and its relation to malignancy, vascularity, and VEGF-A. Clin Cancer Res. 2003 Apr;9(4):1399-405. PMID 12684411
- [Background] Reynes G, Vila V, Martin M, Parada A, Fleitas T, Reganon E, Martinez-Sales V. Circulating markers of angiogenesis, inflammation, and coagulation in patients with glioblastoma. J Neurooncol. 2011 Mar;102(1):35-41. doi: 10.1007/s11060-010-0290-x. Epub 2010 Jul 6. PMID 20607353